CLINICAL TRIAL: NCT06183983
Title: Hitting the Mark: Introducing State-of-the-art MRI for Precision Radiotherapy of Glioblastoma
Acronym: MOSAIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, Radiation oncologist and Associate professor - Department of Radiotherapy, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL84994.078.23
Record Dates: First submitted 2023-12-12; First posted 2023-12-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extended MRI group (Other): In this group, patients with a glioblastoma undergo an extended MRI-scan prior to radiotherapy.
  Interventions: Diagnostic Test: Extended or additional MRI-scan (with contrast) prior to radiotherapy

INTERVENTIONS:
Diagnostic Test: Extended or additional MRI-scan (with contrast) prior to radiotherapy — The MRI-protocol before radiotherapy is extended with 20 minutes. Patients who would not have received an MRI-scan prior to radiotherapy, will get an extra MRI-scan when participating.

SUMMARY:
The goal of this prospective cohort study is to assess the potential of advanced MRI for improved radiotherapy target delineation in patients diagnosed with glioblastoma. The main questions it aims to answer are:

* How does the coverage of the recurrence volume by a radiotherapy plan based on advanced MRI compare to the coverage by the clinical radiotherapy plan?
* How does the distribution of the dose to organs at risk by a radiotherapy plan based on advanced MRI compare to the distribution by the clinical radiotherapy plan?

Participants will undergo an extended MRI-protocol prior to radiotherapy. This extended MRI-protocol includes the clinical brain tumor imaging protocol plus additional advanced MRI-sequences. Radiation treatment and patient follow-up will occur according to the clinical standard.

DETAILED DESCRIPTION:
Rationale: One of the fundamentals of glioblastoma management is radiotherapy, where ionizing radiation is aimed towards a specific target area in the brain to inhibit further tumor growth. As these brain tumors are notorious for their extensive tumor infiltration, where tumor grows beyond the tumor that is visible on conventional magnetic resonance imaging (MRI), this target area, defined as the clinical target volume (CTV), consists of the visible tumor plus a 1.5-cm isotropic safety margin. In the majority of cases, this unspecific CTV margin adequately covers tumor infiltration, but inevitably also includes considerable amounts of healthy tissue. Radiation-induced side-effects like headaches, nausea, fatigue and cognitive decline can substantially affect the quality of life for these patients. An opportunity arises to indirectly visualize tumor infiltration with state-of-the-art advanced MRI (aMRI) techniques, providing additional information on biology rather than only showing anatomical information through conventional MRI. A workflow has been developed to create a CTV based on these aMRI scans (CTVbio) rather than an isotropic expansion. With the additional information that aMRI provides, it could be possible to more accurately define what needs to be targeted and thus minimize damage to healthy tissue. In this research, the aim is to assess the potential of integrating aMRI into radiotherapy target delineation for patients with a glioblastoma by comparing the pattern of failure (coverage of first tumor recurrence by the radiotherapy plan) and the expected radiation dose to organs at risk between the CTVbio and the 1.5-cm CTV. It is hypothesized that the CTVbio can result in decreased radiation dose to organs at risk, whilst having similar pattern of failure.

Primary objective:

• To demonstrate that the probability for reduced coverage of the recurrence volume by a radiotherapy plan based on a CTVbio, compared to the clinical radiotherapy plan (1.5-cm CTV), is lower than 0.20.

Secondary objectives:

* To illustrate a reduction in dose to organs at risk with a radiotherapy plan based on a conceptual CTVbio compared to the clinical radiotherapy plan (1.5-cm CTV).
* To evaluate the synergistic information that each individual aMRI-scan provides for the identification of tumor infiltration.
* To explore the association between pathophysiological changes on aMRI and future tumor recurrence.

Study design: In this prospective cohort study, the clinical standard MRI session used for radiotherapy planning of glioblastoma patients will be extended with aMRI techniques that assess altered oxygenation, angiogenesis and increased protein concentration. In clinical practice at the Erasmus MC, not all patients get an MRI-scan prior to radiotherapy. Patients who would not have received an MRI-scan prior to radiotherapy, will get an extra MRI-scan when they participate in this study. Radiation treatment (and patient follow-up) will occur according to the clinical standard, i.e. using the 1.5-cm CTV for radiotherapy planning. The aMRI-scans will be used to create a theoretical CTVbio and corresponding radiotherapy plan. Pattern-of-failure analysis and assessment of dose to organs at risk will be done to compare the radiotherapy plan based on the 1.5-cm CTV with the (theoretical) radiotherapy plan based on the CTVbio. Additionally, various theoretical CTVs based on different combinations of aMRI-scans are generated to explore the added value of the different aMRI techniques. Lastly, the signal intensities on the aMRI-scans at the site of tumor recurrence are compared with contralateral normal-appearing white matter.

Study population: Patients (≥ 18 years), diagnosed with IDH-wildtype glioblastoma, as confirmed by molecular or immunohistochemistry analysis post resection/biopsy and referred to outpatient clinic of the Department of Radiotherapy to undergo standard treatment with radiotherapy. The inclusion comes to an end when 53 patients have been included.

Intervention: Patients will have an extension to their standard radiotherapy planning MRI-scan taken for regular clinical care (Brain tumor MRI protocol: ± 25 minutes). Patients who would not have received an MRI-scan prior to radiotherapy, will get an extra MRI-scan when they participate in the study. The duration of the extended MRI-scan, which includes the brain tumor MRI protocol, is ± 45 minutes.

Main study parameters/endpoints: Pattern of failure and dose to organs at risk by the radiotherapy plan based on the 1.5-cm CTV and the theoretical plan created with the CTVbio.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: For patients who will already undergo an MRI-scan for radiotherapy, the burden will be an extended MRI-scan (+20 minutes; the total scan time will be 45 minutes instead of 25 minutes). There is no benefit for these patients. For patients who would not have received an MRI-scan prior to radiotherapy, the burden of participation will be an extra MRI-scan (total scan time: 45 minutes) with additional contrast injection. The dosage and administration are similar to the standard Brain tumor MRI protocol, which has often already been acquired before in these patients. The radiation oncologist may decide to use the conventional MRI-scan from this study MRI for target delineation if they believe it has an added value. The use of the conventional MRI-scans is recommended in the ESTRO-EANO guidelines, but is not routinely done for all patients at Erasmus MC. The advanced MRI-scans investigated in this research will not be used by the radiation oncologist

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Adult (18 years or older);
* Diagnosed with IDH-wildtype glioblastoma, as confirmed by pathology including molecular analysis post resection/biopsy;
* Referred to the outpatient clinic of the Dept. of Radiotherapy to undergo standard treatment with radiotherapy (30x2 Gy or 15x2.67Gy or 10x3.4Gy).

Exclusion Criteria:

* Contraindication for (3 Tesla) MRI;
* Contraindication for use of gadolinium-based contrast agent (e.g. subject having renal deficiency or known allergy);
* Referred for treatment of recurrent glioblastoma;
* Previous radiotherapy to the brain;
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pattern-of-failure analysis | The time frame is until tumor recurrence occurs (follow-up for this study will last 2 years maximum for a participant).
  The primary outcome measure is a comparison of the pattern-of-failure by the radiotherapy plan based on CTVbio and the clinical radiotherapy plan (1.5-cm CTV). For both the clinical radiotherapy plan and the aMRI radiotherapy plan of each patient, the recurrence volumes will be classified as in-field, marginal, or distant recurrence if more than 80%, 20-80%, or less than 20% of the recurrence volume falls within the 95% isodose line, respectively.

SECONDARY OUTCOMES:
Distribution of dose to organs at risk. | Through study completion (on average 1 year after the extended MRI-scan).
  The difference in expected dose to important organs at risk between the clinical radiotherapy plan (1.5-cm CTV) and the aMRI radiotherapy plan (CTVbio). Important organs at risk include the brainstem, optic nerves, eyes, lenses, cochlea and optic chiasm.
Recurrence coverage by different combinations of CTVbio | The time frame is until tumor recurrence occurs (follow-up for this study will last 2 years maximum for a participant).
  The differences in tumor recurrence coverage and size between the CTVbio (based on all three aMRI-scans) and CTVs based on individual or other combinations of aMRI, i.e. based on two or one aMRI-scan(s).
Signal intensity on aMRI at the site of tumor recurrence | The time frame is until tumor recurrence occurs (follow-up for this study will last 2 years maximum for a participant).
  The difference in mean and maximum signal intensity on the individual aMRI-scans between the tumor recurrence site and the contralateral normal-appearing white matter.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Méndez Romero, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not available yet